CLINICAL TRIAL: NCT00004175
Title: Phase II Study of Taxotere, Doxorubicin and Cyclophosphamide (TAC) Primary Therapy in Stage III Breast Cancer
Brief Title: Docetaxel, Doxorubicin, and Cyclophosphamide in Treating Women With Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 98B1; NU-98B1; NCI-G99-1643
Record Dates: First submitted 1999-12-10; First posted 2004-03-03 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining docetaxel, doxorubicin, and cyclophosphamide in treating women who have previously untreated stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical response rate to docetaxel, doxorubicin, and cyclophosphamide as primary therapy in women with stage III breast cancer. II. Determine the pathologic complete response rate to this treatment regimen in this patient population. III. Assess the side effects and toxicity profile of this treatment regimen in these patients.

OUTLINE: This is an open label, multicenter study. Patients receive doxorubicin IV over 5-10 minutes followed by cyclophosphamide IV over 5-10 minutes and docetaxel IV over 1 hour. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Within 5 weeks following completion of chemotherapy, operable patients achieving complete or partial response undergo mastectomy, segmental mastectomy, or lumpectomy with nodal dissection. Patients with positive surgical tumor margins may undergo an additional surgical procedure. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed previously untreated, stage III adenocarcinoma of the breast At least one bidimensionally and/or unidimensionally measurable lesion No evidence of disease outside the breast or chest wall, except for ipsilateral axillary lymph nodes Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT no greater than 3 times ULN Alkaline phosphatase no greater than 5 times ULN No acute hepatitis Renal: Creatinine no greater than 1.5 mg/dL No uncontrolled hypercalcemia Cardiovascular: No congestive heart failure LVEF normal No angina pectoris No uncontrolled cardiac arrhythmias No other significant heart disease No myocardial infarction within the past year No superior vena cava syndrome No deep vein thrombosis requiring anticoagulant therapy Neurologic: No dementia No seizures No concurrent grade 2 or greater peripheral neuropathy Other: No medical instability No active infection No gastrointestinal bleeding No uncontrolled diabetes No psychological, familial, sociological, or geographical conditions or other circumstances that would preclude study No other malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix No history of hypersensitivity to polysorbate 80 Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy for breast cancer Chemotherapy: No prior chemotherapy for breast cancer Endocrine therapy: No prior hormonal therapy for breast cancer No concurrent corticosteroids except for chronic methylprednisolone or equivalent for more than 6 months duration at no more than 20 mg/day Radiotherapy: Not specified Surgery: Not specified Other: At least 3 weeks since prior investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Primary Completion 2004-09 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (4):
- United States (4):
  - Stanford University Medical Center, Stanford, California
  - Monroe Medical Associates, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York